CLINICAL TRIAL: NCT02805426
Title: Double-blind, Randomized Controlled Trial to Assess the Effectiveness of Tranexamic Acid When Used as an Adjunct to Misoprostol for the Treatment of Postpartum Hemorrhage
Brief Title: Effectiveness of Tranexamic Acid When Used as an Adjunct to Misoprostol for the Treatment of Postpartum Hemorrhage
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Gynuity Health Projects (Other)
Collaborators: Center for Research and Consultancy in Reproductive Health (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 3006
Record Dates: First submitted 2016-03-09; First posted 2016-06-20 (Estimated); Last update posted 2018-02-19 (Actual); Status verified 2018-02

CONDITIONS: Postpartum Hemorrhage
MeSH Terms: conditions — Postpartum Hemorrhage | interventions — Tranexamic Acid; Misoprostol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Tranexamic acid (Experimental): 1950 mg oral tranexamic acid + 800 mcg sublingual misoprostol
  Interventions: Drug: Tranexamic Acid; Drug: Misoprostol
- Placebo (Placebo Comparator): oral placebo + 800 mcg sublingual misoprostol
  Interventions: Drug: Placebo; Drug: Misoprostol

INTERVENTIONS:
Drug: Tranexamic Acid
  Arms: Tranexamic acid
Drug: Placebo
  Arms: Placebo
Drug: Misoprostol

SUMMARY:
This study is a randomized, double-blind, placebo controlled trial that will enroll 250 women (125 per study arm).

The objective of the study is to determine the efficacy and tolerability of oral tranexamic acid when used as an adjunct to misoprostol for treatment of postpartum hemorrhage (PPH). Women will be diagnosed with postpartum hemorrhage if blood loss reaches 700ml in the calibrated receptacle. If diagnosed with postpartum hemorrhage , the woman will be randomized to receive either tranexamic acid or placebo, both in tablet form. All participants will receive 800 mcg sublingual misoprostol (4 tablets 200mcg each).

The investigators hypothesize that tranexamic acid (in tablet form) as an adjunct to misoprostol will be more effective than misoprostol alone in stopping postpartum bleeding without recourse to further treatment in significantly more women.

ELIGIBILITY:
Inclusion Criteria:

* Women who delivery vaginally
* Women who experience PPH defined as blood loss ≥700ml
* Women capable of giving consent

Exclusion Criteria:

* Clear contraindication for tranexamic acid such as known allergy or thromboembolic event during pregnancy
* Women delivering via cesarean section
* Provider feels that the woman, at presentation for delivery, is not in a position to give appropriate informed consent

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 260 (Actual)
Dates: Start 2016-10; Primary Completion 2018-01 (Actual); Study Completion 2018-01 (Actual)

PRIMARY OUTCOMES:
Proportion of women with bleeding controlled with the study regimens alone, without recourse to further treatment in each study arm | 20 minutes after initial study treatment

SECONDARY OUTCOMES:
Rate of severe PPH | 2 hours after delivery
  Rate of severe PPH (>1000 ml total blood loss)
Mean/median blood loss | at two hours after treatment
Proportion of women with controlled bleeding | At various time intervals after study treatment (20, 40, 60, 120 mins)
  proportion of women with bleeding controlled at different time intervals (20, 40, 60, 120 mins)
Use of uterotonic agents after initial treatment | 2 hours after delivery
  Proportion of women who are given uterotonic agents after initial treatment
Proportion of women who received a serious interventions | 2 hours after delivery
  Serious intervention is defined as blood transfusion, interventions for tissue repair, surgical intervention [including curettage, vacuum aspiration for retained placental tissue, hysterectomy, surgical uterine artery ligature])
Proportion of women who received additional drugs | 2 hours after delivery
  Proportion of women who receive additional drugs
Proportion of women who receive additional intervention | 2 hours after delivery
  Proportion of women who receive additional interventions (i.e. suturing)
Adverse events | 48 hours after delivery
  Proportion of women who experience an adverse event
Proportion of women who experience side effects | 2 hours after delivery
  Proportion of women who experience side effects
Proportion of women who find the treatment tolerable | 48 hours after delivery
  Proportion of women who find the procedure tolerable and acceptable as indicated in an acceptability scale

CONTACTS AND LOCATIONS:
Overall Officials: Beverly Winikoff, MD, MPH, Principal Investigator — Gynuity Health Projects; Jill Durocher, Principal Investigator — Gynuity Health Projects; Dina Abbas, MPH, Principal Investigator — Gynuity Health Projects; Nguyen thi Nhu Ngoc, MD, MSc, Principal Investigator — CRCRH; Ayisha Diop, MPH, Principal Investigator — Gynuity Health Projects
Locations (4):
- Senegal (2):
  - Centre de santé 10ème de Thiès, Thiès
  - Centre hospitalier Régional de Thiès, Ahmadou Sakhir Ndiéguène, Thiès
- Vietnam (2):
  - National OB-GYN Hospital, Hanoi
  - Hung Vuong Hospital, Ho Chi Minh City

REFERENCES:
- [Derived] Diop A, Abbas D, Ngoc NTN, Martin R, Razafi A, Tuyet HTD, Winikoff B. A double-blind, randomized controlled trial to explore oral tranexamic acid as adjunct for the treatment for postpartum hemorrhage. Reprod Health. 2020 Mar 6;17(1):34. doi: 10.1186/s12978-020-0887-2. PMID 32143721